CLINICAL TRIAL: NCT00236899
Title: A Randomized Phase III Trial of Gemcitabine and Docetaxel Versus Gemcitabine and Paclitaxel in Patients With Metastatic Breast Cancer: A Comparison of Different Schedules
Brief Title: Phase III Study of Two Different Schedules (Weekly and Tri-weekly) of Combination of Gemcitabine and Two Taxanes in MBC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 9846; B9E-IT-S376 (Other: Eli Lilly and Company)
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Results first posted 2011-09-27 (Estimated); Last update posted 2011-09-27 (Estimated); Status verified 2011-08

CONDITIONS: Metastatic Breast Cancer (MBC)
MeSH Terms: conditions — Breast Neoplasms | interventions — Gemcitabine; Docetaxel; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- A: Docetaxel and Gemcitabine (Tri-weekly) (Experimental): Docetaxel and Gemcitabine (Tri-weekly)
  Interventions: Drug: Gemcitabine; Drug: Docetaxel
- B: Paclitaxel and Gemcitabine (Tri-weekly) (Experimental): Paclitaxel and Gemcitabine (Tri-weekly)
  Interventions: Drug: Gemcitabine; Drug: Paclitaxel
- C: Docetaxel and Gemcitabine (Weekly) (Experimental): Docetaxel and Gemcitabine (Weekly)
  Interventions: Drug: Gemcitabine; Drug: Docetaxel
- D: Paclitaxel and Gemcitabine (Weekly) (Experimental): Paclitaxel and Gemcitabine (Weekly)
  Interventions: Drug: Gemcitabine; Drug: Paclitaxel

INTERVENTIONS:
Drug: Gemcitabine — Arm A: 1000 mg/m², 30 minute (min) intravenous (IV) infusion on Days 1 and 8, repeated every 21 days for 10 cycles for complete responders (CRs=disappearance of all target lesions) or partial responders (PRs≥30% decrease in sum of longest diameter of target lesions); 6 cycles for stable disease (SD=small changes that do not meet the above criteria); or until progressive disease (PD≥20% increase in sum of longest diameter of target lesions).
  Arm B: 1250 mg/m², 30 min IV infusion on Days 1 and 8, repeated every 21 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Arm C: 800 mg/m², 30 min IV infusion on Days 1, 8, and 15 repeated every 21 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Arm D: 800 mg/m², 30 min IV infusion on Days 1, 8, and 15 repeated every 28 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Other Names: LY188011; Gemzar
Drug: Docetaxel — Arm A: 75 milligram per square meter (mg/m²), 60 min IV infusion on Day 1 only, to be given 30 min prior to Gemcitabine, repeated every 21 days (tri-weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Arm C: 30 mg/m², 30-60 min IV infusion on Days 1, 8, and 15, to be given 30 min prior to Gemcitabine, repeated every 28 days (weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Arms: A: Docetaxel and Gemcitabine (Tri-weekly); C: Docetaxel and Gemcitabine (Weekly)
Drug: Paclitaxel — Arm B: 175 mg/m², IV infusion over approximately 3 hours, followed by Gemcitabine, on Day 1, repeated every 21 days (tri-weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Arm D: 80 mg/m², IV infusion over approximately 1 hour, Days 1, 8, and 15, followed by Gemcitabine, repeated every 28 days (weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Arms: B: Paclitaxel and Gemcitabine (Tri-weekly); D: Paclitaxel and Gemcitabine (Weekly)

SUMMARY:
Multi-center, randomized Phase III study. 4 arms. 360 Patient to enroll. Purpose is evaluate time to progression disease (PD).

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of metastatic breast cancer (MBC).
* Prior neoadjuvant or adjuvant taxanes regimen is allowed if ≥12 months since completion of the regimen.
* Relapsing after receiving one adjuvant/neoadjuvant chemotherapy containing an anthracycline if not clinically contraindicated.
* Patients with measurable disease.
* Previous hormonal therapy for adjuvant setting or metastatic disease.

Exclusion Criteria:

* Previous chemotherapy for MBC
* Previous chemotherapy with gemcitabine in any setting of disease
* Patient candidable to treatment with trastuzumab.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 241 (Actual)
Dates: Start 2005-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon-Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Chair — Eli Lilly and Company
Locations (34):
- Italy (34):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Avellino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bologna
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brescia
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cagliari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Candiolo-Torino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Casale Monferrato
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Castelfranco Veneto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Catania
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cuneo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ferrara
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Frosinone
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Genova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gorgonzola
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lecce
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mantova
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Milan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Napoli
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Negrar
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Padua
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Parma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Piacenza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pisa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Potenza
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Reggio Calabria
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rome
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Sisto
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sassari
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Taormina
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Torino
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trento
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Treviglio
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Trieste
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Udine
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Viterbo

REFERENCES:
- [Derived] Del Mastro L, Fabi A, Mansutti M, De Laurentiis M, Durando A, Merlo DF, Bruzzi P, La Torre I, Ceccarelli M, Kazeem G, Marchi P, Boy D, Venturini M, De Placido S, Cognetti F. Randomised phase 3 open-label trial of first-line treatment with gemcitabine in association with docetaxel or paclitaxel in women with metastatic breast cancer: a comparison of different schedules and treatments. BMC Cancer. 2013 Mar 28;13:164. doi: 10.1186/1471-2407-13-164. PMID 23537313
- See also: Lilly Clinical Trial Registry — http://www.lillytrials.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Docetaxel and Gemcitabine (Tri-weekly): Docetaxel: 75 milligram per square meter (mg/m²), 60 minute (min) intravenous (IV) infusion on Day 1 only, to be given 30 min prior to Gemcitabine, repeated every 21 days (tri-weekly) for 10 cycles for complete responders (CRs=disappearance of all target lesions) or partial responders (PRs≥30% decrease in sum of longest diameter of target lesions); 6 cycles for stable disease (SD=small changes that do not meet the above criteria); or until progressive disease (PD≥20% increase in sum of longest diameter of target lesions).
  Gemcitabine: 1000 mg/m², 30 min IV infusion on Days 1 and 8, repeated every 21 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
- Arm B: Paclitaxel and Gemcitabine (Tri-weekly): Paclitaxel: 175 mg/m², IV infusion over approximately 3 hours followed by Gemcitabine on Day 1, repeated every 21 days (tri-weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Gemcitabine: 1250 mg/m², 30 min IV infusion on Days 1 and 8, repeated every 21 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
- Arm C: Docetaxel and Gemcitabine (Weekly): Docetaxel: 30 mg/m², 30-60 min IV infusion on Days 1, 8, and 15 to be given 30 minutes prior Gemcitabine, repeated every 28 days (weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Gemcitabine: 800 mg/m², 30 min IV infusion on Days 1, 8, and 15 repeated every 28 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
- Arm D: Paclitaxel and Gemcitabine (Weekly): Paclitaxel: 80 mg/m², IV infusion over approximately 1 hour, Days 1, 8, and 15, followed by Gemcitabine, repeated every 28 days (weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Gemcitabine: 800 mg/m², 30 min IV infusion on Days 1, 8, and 15 repeated every 28 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
Period: Overall Study
Arm/Group | Arm A: Docetaxel and Gemcitabine (Tri-weekly) | Arm B: Paclitaxel and Gemcitabine (Tri-weekly) | Arm C: Docetaxel and Gemcitabine (Weekly) | Arm D: Paclitaxel and Gemcitabine (Weekly)
Started | 60 | 64 | 58 | 59
Completed | 18 | 24 | 14 | 19
Not Completed | 42 | 40 | 44 | 40
Not completed — Adverse Event (Study Related) | 1 | 1 | 2 | 1
Not completed — Adverse Event (Not Study Related) | 3 | 3 | 4 | 7
Not completed — Death (Study Disease) | 1 | 4 | 0 | 0
Not completed — Death (Not Study Related) | 2 | 0 | 0 | 0
Not completed — Death (Study Drug Toxicity) | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0
Not completed — Entry Criteria Exclusion | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 6 | 4 | 5 | 2
Not completed — Physician Decision | 7 | 8 | 7 | 6
Not completed — Satisfactory Response | 2 | 0 | 0 | 1
Not completed — Lack of Efficacy | 18 | 18 | 25 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Docetaxel and Gemcitabine (Tri-weekly) | Arm B: Paclitaxel and Gemcitabine (Tri-weekly) | Arm C: Docetaxel and Gemcitabine (Weekly) | Arm D: Paclitaxel and Gemcitabine (Weekly) | Total
Number analyzed (Participants) | 60 | 64 | 58 | 59 | 241
Age Continuous [Mean (Standard Deviation); unit: years] | 56.58 (10.21) | 56.31 (9.84) | 55.78 (8.99) | 54.66 (10.04) | 55.85 (9.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 64 | 58 | 59 | 241
  Male | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 58 | 63 | 58 | 59 | 238
  Other | 2 | 1 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Italy | 60 | 64 | 58 | 59 | 241
Menopausal Status [Number; unit: participants] — Menopausal status is defined as the number of participants with premenopausal or postmenopausal status.
  participants
    Premenopausal | 19 | 17 | 16 | 21 | 73
    Postmenopausal | 41 | 47 | 42 | 38 | 168
Previous Hormonal Therapy [Number; unit: participants] — Previous hormonal therapy status is defined as the number of participants who had previously received hormonal therapy.
  participants
    Yes | 44 | 48 | 40 | 46 | 178
    No | 16 | 16 | 17 | 13 | 62
    Unknown | 0 | 0 | 1 | 0 | 1
Presence or Absence of Visceral Metastases [Number; unit: participants] — Visceral metastases are defined as any metastases to the major organs excluding bone, skin, soft tissue, and lymph nodes.
  participants
    Absence | 19 | 19 | 16 | 23 | 77
    Presence | 41 | 45 | 42 | 36 | 164
Number of Participants with Previous Adjuvant/Neoadjuvant Taxane Therapy [Number; unit: participants] — This baseline measure presents the number of participants who had previously received adjuvant/neoadjuvant taxane therapy.
  participants
    Yes | 21 | 24 | 12 | 19 | 76
    No | 39 | 40 | 45 | 40 | 164
    Unknown | 0 | 0 | 1 | 0 | 1
Quality of Life (QOL) using the Rotterdam Symptom Scale Checklist (RSSC) [Number; unit: participants] — The RSSC is a valid and reliable instrument use to measure psychological and physical distress of cancer patients. The overall QOL of patients are assessed and categorized as: Excellent, Good, Moderately Good, Neither Good nor Bad, Rather Poor, Poor, and Extremely Poor.
  participants
    Excellent | 5 | 2 | 2 | 1 | 10
    Good | 17 | 15 | 14 | 13 | 59
    Moderately Good | 6 | 10 | 7 | 10 | 33
    Neither Good Nor Bad | 8 | 6 | 6 | 8 | 28
    Rather Poor | 6 | 4 | 1 | 8 | 19
    Poor | 1 | 2 | 5 | 3 | 11
    Extremely Poor | 2 | 1 | 1 | 0 | 4
    No Response | 15 | 24 | 22 | 16 | 77

OUTCOME MEASURES:

1. Primary Outcome: Time to Progressive Disease (TTPD) by Treatment Schedule
Description: TTPD is defined as the time from the day of treatment to first observation of documented disease progression or death due to any cause, whichever comes first. TTPD was censored at the time of last follow-up for patients who were still alive without progression. Tumor response was assessed in cancer patients by using Response Evaluation Criteria in Solid Tumors (RECIST), which define when cancer patients improve ("respond"), stay the same ("stabilize"), or worsen ("progression") during treatments. Progressive Disease is a ≥20% increase in sum of longest diameter of target lesions.
Time Frame: Baseline up to 49.84 months
Population: Intention to treat (ITT) population is defined as the population of all randomized participants. Treatment arms based on treatment schedule (Weekly vs 3 Weekly) were combined for this population. A total of 33 participants were censored with 16 (13.68%)in the Weekly arm and 17 (13.71%) participants in the 3 Weekly arm.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Treatment Schedule (Weekly): Arm C, Docetaxel and Gemcitabine (Weekly):
  Docetaxel: 30 mg/m², 30-60 min IV infusion on Days 1, 8, and 15 to be given 30 minutes prior to Gemcitabine, repeated every 28 days (weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Gemcitabine: 800 mg/m², 30 min IV infusion on Days 1, 8, and 15 repeated every 28 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Arm D, Paclitaxel and Gemcitabine (Weekly):
  Paclitaxel: 80 mg/m², IV infusion over approximately 1 hour, Days 1, 8, and 15, followed by Gemcitabine, repeated every 28 days (weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Gemcitabine: 800 mg/m², 30 min IV infusion on Days 1, 8, and 15 repeated every 28 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
- Treatment Schedule (3 Weekly): Arm A, Docetaxel and Gemcitabine (3 Weekly):
  Docetaxel: 75 mg/m², 60 min IV infusion on Day 1 only, to be given 30 min prior to Gemcitabine, repeated every 21 days (tri-weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Gemcitabine: 1000 mg/m², 30 min IV infusion on Days 1 and 8, repeated every 21 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Arm B, Paclitaxel and Gemcitabine (3 Weekly):
  Paclitaxel: 175 mg/m², IV infusion over approximately 3 hours followed by Gemcitabine, repeated every 21 days (tri-weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Gemcitabine: 1250 mg/m², 30 min IV infusion on Days 1 and 8, repeated every 21 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
Arm/Group | Treatment Schedule (Weekly) | Treatment Schedule (3 Weekly)
Number analyzed (Participants) | 117 | 124
months | 8.33 [6.19 to 10.16] | 7.51 [5.93 to 8.33]
Statistical Analysis 1: Comparison: Treatment Schedule (Weekly) vs Treatment Schedule (3 Weekly); Test type: Superiority or Other; p = 0.345, Regression, Cox; Hazard Ratio (HR) = 1.14, 95% CI [0.87 to 1.50]

2. Secondary Outcome: Overall Survival (OS) by Treatment Schedule
Description: OS is the duration from enrollment to time of death as a result of any cause. For participants who are alive, OS is censored at the last contact (date of the last follow-up visit).
Time Frame: Baseline up to 51.64 months
Population: Intention to treat (ITT) population defined as the population of all randomized participants. Treatment arms based on treatment schedule (Weekly vs 3 Weekly) were combined for this population. A total of 109 (45.2%) participants were censored with 53 (45.3%) in the Weekly arm and 56 (45.2%) participants in the 3 Weekly arm.
Measure: Mean (95% Confidence Interval); unit: months
Arm/Group | Treatment Schedule (Weekly) | Treatment Schedule (3 Weekly)
Number analyzed (Participants) | 117 | 124
months | 21.11 [17.28 to 26.75] | 20.95 [18.92 to 33.21]
Statistical Analysis 1: Comparison: Treatment Schedule (Weekly) vs Treatment Schedule (3 Weekly); Test type: Superiority or Other; p = 0.885, Regression, Cox; Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.69 to 1.37]

3. Secondary Outcome: Overall Survival (OS) by Treatment Drug
Description: as for outcome 2
Time Frame: Baseline up to 51.64 months
Population: ITT population defined as the population of all randomized participants. Treatment arms based on Treatment Drug (Docetaxel+Gemcitabine vs Paclitaxel+Gemcitabine) were combined for this population. A total of 109 participants were censored with 55 (46.61%) in the Docetaxel+Gemcitabine arm and 54 (43.90%) in the Paclitaxel+Gemcitabine arm.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Treatment Drug (Docetaxel): Arm A, Docetaxel: 75 mg/m², 60 min IV infusion on Day 1 only, to be given 30 min prior to Gemcitabine, repeated every 21 days (tri-weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Gemcitabine: 1000 mg/m² 30 min IV infusion on Days 1 and 8, repeated every 21 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Arm C, Docetaxel: 30 mg/m², 30-60 min IV infusion on Days 1, 8, and 15 to be given 30 min prior to Gemcitabine, repeated every 28 days (weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Gemcitabine: 800 mg/m², 30 min IV infusion on Days 1, 8, and 15, repeated every 28 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
- Treatment Drug (Paclitaxel): Arm B, Paclitaxel: 175 mg/m², IV infusion over approximately 3 hours followed by followed by Gemcitabine on Day 1, repeated every 21 days (tri-weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Gemcitabine: 1250 mg/m², 30 min IV infusion on Days 1 and 8, repeated every 21 days (tri-weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Arm D, Paclitaxel: 80 mg/m², IV infusion over approximately 1 hour, Days 1, 8, and 15 followed by Gemcitabine, repeated every 28 days (weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Gemcitabine: 800 mg/m², 30 min IV infusion on Days 1, 8, and 15 repeated every 28 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until disease progression.
Arm/Group | Treatment Drug (Docetaxel) | Treatment Drug (Paclitaxel)
Number analyzed (Participants) | 118 | 123
months | 19.11 [16.59 to 24.00] | 23.80 [19.38 to 31.97]
Statistical Analysis 1: Comparison: Treatment Drug (Docetaxel) vs Treatment Drug (Paclitaxel); Test type: Superiority or Other; p = 0.976, Regression, Cox; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.71 to 1.42]

4. Secondary Outcome: Overall Response Rate (ORR) by Treatment Schedule
Description: Response using Response Evaluation Criteria In Solid Tumors (RECIST) criteria. Complete Response=disappearance of all target lesions; Partial Response≥30% decrease in sum of longest diameter of target lesions; Progressive Disease≥20% increase in sum of longest diameter of target lesions; Stable Disease=small changes that do not meet above criteria. Not Available=participants assessed whose data were not available. Not Assessed=participants who did not participate in assessments. The ORR=sum of complete and partial tumor responses observed, divided by the total number of evaluable participants.
Time Frame: Baseline up to 49.84 months
Population: All randomized patients treated with at least 1 dose of Docetaxel, Paclitaxel or Gemcitabine. Treatment arms based on treatment schedule (Weekly vs 3 Weekly) were combined for this population.
Measure: Number; unit: percentage of responses
Arm/Group | Treatment Schedule (Weekly) | Treatment Schedule (3 Weekly)
Number analyzed (Participants) | 117 | 124
percentage of responses
  ORR (Complete Response or Partial Response) | 50.43 | 33.06
  Complete Response | 6.84 | 5.65
  Partial Response | 43.59 | 27.42
  Stable Disease | 23.93 | 40.32
  Progressive Disease | 21.37 | 12.90
  Not Available | 0.85 | 1.61
  Not Assessed | 3.42 | 12.10
Statistical Analysis 1: Comparison: Treatment Schedule (Weekly) vs Treatment Schedule (3 Weekly); Test type: Superiority or Other; p = 0.0028, Regression, Logistic; Odds Ratio (OR) = 0.442, 95% CI 2-sided [0.259 to 0.754]

5. Primary Outcome: Time to Progressive Disease (TTPD) by Treatment Drug
Description: as for outcome 1
Time Frame: Baseline up to 49.84 months
Population: ITT population defined as the population of all randomized participants. Treatment arms based on Treatment Drug (Docetaxel+Gemcitabine vs Paclitaxel+Gemcitabine) were combined for this population. A total of 33 (13.7%) participants were censored with 17 (13.68%) in the Docetaxel+Gemcitabine arm and 18 (13.71%) in the Paclitaxel+Gemcitabine arm.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Drug (Docetaxel) | Treatment Drug (Paclitaxel)
Number analyzed (Participants) | 118 | 123
months | 7.74 [5.57 to 9.80] | 7.80 [6.20 to 8.72]
Statistical Analysis 1: Comparison: Treatment Drug (Docetaxel) vs Treatment Drug (Paclitaxel); Test type: Superiority or Other; p = 0.150, Regression, Cox; Hazard Ratio (HR) = 1.23, 95% CI 2-sided [0.93 to 1.62]

6. Secondary Outcome: Overall Response Rate(ORR) by Treatment Drug
Description: as for outcome 4
Time Frame: Baseline up to 49.84 months
Population: All randomized participants treated with at least 1 dose of Docetaxel, Paclitaxel or Gemcitabine. Treatment arms based on Treatment Drug (Docetaxel+Gemcitabine vs Paclitaxel+Gemcitabine) were combined for this population.
Measure: Number; unit: percentage of responses
Arm/Group | Treatment Drug (Docetaxel) | Treatment Drug (Paclitaxel)
Number analyzed (Participants) | 118 | 123
percentage of responses
  ORR (Complete Response or Partial Response) | 43.2 | 39.8
  Complete Response | 5.08 | 7.32
  Partial Response | 38.14 | 32.52
  Stable Disease | 32.20 | 32.52
  Progressive Disease | 17.80 | 16.26
  Not Available | 0.85 | 1.63
  Not Assessed | 5.93 | 9.76
Statistical Analysis 1: Comparison: Treatment Drug (Docetaxel) vs Treatment Drug (Paclitaxel); Test type: Superiority or Other; p = 0.4567, Regression, Logistic; Odds Ratio (OR) = 0.818, 95% CI 2-sided [0.482 to 1.389]

7. Secondary Outcome: Number of Participants With Serious and Nonserious Adverse Events (AEs)
Description: Summary tables of serious adverse events (SAEs) and all other nonserious AEs are located in the Reported Adverse Event Module.
Time Frame: Baseline up to 51.64 months
Population: Intent to treat (ITT) population defined as the population of all randomized participants.
Measure: Number; unit: participants
Groups:
- Arm A: Docetaxel and Gemcitabine (Tri-weekly): Docetaxel: 75 milligram per square millimeter (mg/m²), 60 minute (min) intravenous (IV) infusion on Day 1 only, to be given 30 min prior to Gemcitabine, repeated every 21 days (tri-weekly) for 10 cycles for complete responders (CRs=disappearance of all target lesions) or partial responders (PRs=≥30% decrease in sum of longest diameter of target lesions); 6 cycles for stable disease (SD=small changes that do not meet the above criteria); or until progressive disease (PD≥20% increase in sum of longest diameter of target lesions).
  Gemcitabine: 1000 mg/m², 30 min IV infusion on Days 1 and 8, repeated every 21 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
- Arm B: Paclitaxel and Gemcitabine (Tri-weekly): Paclitaxel: 175 mg/m², IV infusion over approximately 3 hours followed by Gemcitabine, repeated every 21 days (tri-weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Gemcitabine: 1250 mg/m², 30 min IV infusion on Days 1 and 8, repeated every 21 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
- Arm C: Docetaxel and Gemcitabine (Weekly): Docetaxel: 30 mg/m², 30-60 min IV infusion on Days 1, 8, and 15 to be given 30 minutes prior to Gemcitabine, repeated every 28 days (weekly) for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
  Gemcitabine: 800 mg/m², 30 min IV infusion on Days 1, 8, and 15 repeated every 28 days for 10 cycles for CRs or PRs; 6 cycles for SD; or until PD.
Arm/Group | Arm A: Docetaxel and Gemcitabine (Tri-weekly) | Arm B: Paclitaxel and Gemcitabine (Tri-weekly) | Arm C: Docetaxel and Gemcitabine (Weekly) | Arm D: Paclitaxel and Gemcitabine (Weekly)
Number analyzed (Participants) | 59 | 62 | 58 | 59
participants
  SAEs | 9 | 10 | 7 | 11
  Nonserious AEs | 57 | 58 | 53 | 56

8. Secondary Outcome: Quality of Life (QOL) Using the Rotterdam Symptom Scale Checklist (RSSC) at Beginning of 3-Week or 4-Week Cycle
Description: RSSC is a valid and reliable measure of psychological and physical distress of cancer patients. Overall QOL is assessed on a 7-point scale (1=Excellent to 7=Extremely Poor). Categories include Excellent, Good, Moderately Good, Neither Good nor Bad, Rather Poor, Poor, and Extremely Poor. Number of responses to the overall QOL by treatment arm are provided. Arms A (Docetaxel and Gemcitabine 3 Weekly) and B (Paclitaxel and Gemcitabine 3 Weekly) were assessed every 3 weeks. Arms C (Docetaxel and Gemcitabine Weekly) and D (Paclitaxel and Gemcitabine Weekly) were assessed every 4 weeks.
Time Frame: Baseline up to 51.64 months
Population: Intent to treat (ITT) population defined as all randomized participants.
Measure: Number; unit: participants
Arm/Group | Arm A: Docetaxel and Gemcitabine (Tri-weekly) | Arm B: Paclitaxel and Gemcitabine (Tri-weekly) | Arm C: Docetaxel and Gemcitabine (Weekly) | Arm D: Paclitaxel and Gemcitabine (Weekly)
Number analyzed (Participants) | 60 | 64 | 58 | 59
participants
  1=Excellent | 3 | 1 | 2 | 4
  2=Good | 13 | 13 | 9 | 5
  3=Moderately Good | 6 | 8 | 9 | 9
  4=Neither Good Nor Bad | 6 | 7 | 6 | 7
  5=Rather Poor | 2 | 3 | 3 | 6
  6=Poor | 0 | 3 | 7 | 2
  7=Extremely Poor | 0 | 3 | 0 | 1
  No Response | 30 | 26 | 22 | 25
Statistical Analysis 1: Comparison: Arm B: Paclitaxel and Gemcitabine (Tri-weekly) vs Arm D: Paclitaxel and Gemcitabine (Weekly); Test type: Superiority or Other; p = 0.142, Fisher Exact — This is the p-value for Treatment Schedule (Docetaxel and Gemcitabine 3 Weekly + Paclitaxel and Gemcitabine 3 Weekly) and Treatment Drug (Docetaxel and Gemcitabine Weekly + Paclitaxel and Gemcitabine Weekly)
Statistical Analysis 2: Comparison: Arm A: Docetaxel and Gemcitabine (Tri-weekly) vs Arm C: Docetaxel and Gemcitabine (Weekly); Test type: Superiority or Other; p = 0.470, Fisher Exact — This is the p-value for Treatment Drug (Docetaxel and Gemcitabine 3 Weekly + Docetaxel and Gemcitabine Weekly vs Paclitaxel and Gemcitabine 3 Weekly + Paclitaxel and Gemcitabine Weekly)

9. Secondary Outcome: Quality of Life (QOL) Using the Rotterdam Symptom Scale Checklist (RSSC) at 30-Day Post-therapy Visit
Description: RSSC is a valid and reliable measure of psychological and physical distress of cancer patients. Overall QOL is assessed on a 7-point scale (1=Excellent to 7=Extremely Poor). Categories include Excellent, Good, Moderately Good, Neither Good nor Bad, Rather Poor, Poor, and Extremely Poor. Number of responses to the overall QOL (using the 7-point scale) by treatment arm are provided.
Time Frame: Baseline up to 51.64 months
Population: Intent to treat (ITT) population defined as all randomized participants.
Measure: Number; unit: participants
Arm/Group | Arm A: Docetaxel and Gemcitabine (Tri-weekly) | Arm B: Paclitaxel and Gemcitabine (Tri-weekly) | Arm C: Docetaxel and Gemcitabine (Weekly) | Arm D: Paclitaxel and Gemcitabine (Weekly)
Number analyzed (Participants) | 60 | 64 | 58 | 59
participants
  1=Excellent | 0 | 0 | 0 | 0
  2=Good | 7 | 7 | 2 | 4
  3=Moderately Good | 2 | 6 | 3 | 2
  4=Neither Good Nor Bad | 3 | 6 | 0 | 3
  5=Rather Poor | 0 | 1 | 1 | 1
  6=Poor | 2 | 0 | 1 | 2
  7=Extremely Poor | 1 | 0 | 2 | 0
  No Response | 45 | 44 | 49 | 47
Statistical Analysis 1: Comparison: Arm B: Paclitaxel and Gemcitabine (Tri-weekly) vs Arm D: Paclitaxel and Gemcitabine (Weekly); Test type: Superiority or Other; p = 0.293, Fisher Exact — [p-value comment as in outcome 8, analysis 1]
Statistical Analysis 2: Comparison: Arm A: Docetaxel and Gemcitabine (Tri-weekly) vs Arm C: Docetaxel and Gemcitabine (Weekly); Test type: Superiority or Other; p = 0.476, Fisher Exact — [p-value comment as in outcome 8, analysis 2]

ADVERSE EVENTS:
Arm/Group | Arm A: Docetaxel and Gemcitabine (Tri-weekly) | Arm B: Paclitaxel and Gemcitabine (Tri-weekly) | Arm C: Docetaxel and Gemcitabine (Weekly) | Arm D: Paclitaxel and Gemcitabine (Weekly)
Serious Adverse Events (participants affected / at risk) | 9/59 | 10/62 | 7/58 | 11/59
Other Adverse Events (participants affected / at risk) | 57/59 | 58/62 | 53/58 | 56/59
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Docetaxel and Gemcitabine (Tri-weekly) (N=59) | Arm B: Paclitaxel and Gemcitabine (Tri-weekly) (N=62) | Arm C: Docetaxel and Gemcitabine (Weekly) (N=58) | Arm D: Paclitaxel and Gemcitabine (Weekly) (N=59)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Meningitis pneumococcal (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis syndrome (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hydropneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Femoral artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vasculitis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Docetaxel and Gemcitabine (Tri-weekly) (N=59) | Arm B: Paclitaxel and Gemcitabine (Tri-weekly) (N=62) | Arm C: Docetaxel and Gemcitabine (Weekly) (N=58) | Arm D: Paclitaxel and Gemcitabine (Weekly) (N=59)
Anaemia (Blood and lymphatic system disorders) | 12 (19) | 10 (13) | 12 (15) | 17 (23)
Leukopenia (Blood and lymphatic system disorders) | 21 (41) | 9 (15) | 14 (35) | 13 (30)
Lymphopenia (Blood and lymphatic system disorders) | 3 (5) | 2 (3) | 3 (5) | 2 (5)
Neutropenia (Blood and lymphatic system disorders) | 50 (154) | 33 (85) | 20 (71) | 38 (90)
Thrombocytopenia (Blood and lymphatic system disorders) | 4 (4) | 3 (6) | 10 (25) | 12 (19)
Conjunctivitis (Eye disorders) | 1 (1) | 2 (2) | 4 (5) | 4 (5)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 7 (7) | 3 (4) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 5 (5) | 4 (4) | 5 (6) | 1 (1)
Constipation (Gastrointestinal disorders) | 8 (8) | 9 (10) | 10 (16) | 9 (9)
Diarrhoea (Gastrointestinal disorders) | 18 (27) | 11 (13) | 21 (37) | 14 (24)
Gastritis (Gastrointestinal disorders) | 3 (3) | 0 (0) | 2 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 25 (38) | 21 (34) | 20 (34) | 21 (33)
Stomatitis (Gastrointestinal disorders) | 10 (13) | 3 (4) | 8 (10) | 2 (2)
Vomiting (Gastrointestinal disorders) | 13 (18) | 10 (17) | 11 (17) | 4 (6)
Asthenia (General disorders) | 17 (34) | 18 (28) | 18 (40) | 15 (28)
Fatigue (General disorders) | 15 (18) | 12 (16) | 13 (24) | 18 (28)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Mucosal inflammation (General disorders) | 17 (26) | 7 (8) | 10 (11) | 6 (9)
Oedema (General disorders) | 2 (2) | 2 (2) | 6 (7) | 4 (5)
Oedema peripheral (General disorders) | 1 (1) | 2 (3) | 4 (6) | 6 (9)
Pyrexia (General disorders) | 17 (22) | 16 (27) | 23 (32) | 17 (38)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 1 (2) | 0 (0) | 4 (4)
Hypertransaminasaemia (Hepatobiliary disorders) | 4 (5) | 2 (2) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
Alanine aminotransferase increased (Investigations) | 11 (18) | 14 (28) | 17 (46) | 20 (30)
Aspartate aminotransferase increased (Investigations) | 8 (10) | 12 (13) | 12 (25) | 13 (21)
Blood alkaline phosphatase increased (Investigations) | 3 (5) | 1 (1) | 3 (4) | 3 (3)
Blood lactate dehydrogenase increased (Investigations) | 1 (2) | 0 (0) | 0 (0) | 3 (4)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 4 (4) | 3 (4) | 4 (5)
Haemoglobin decreased (Investigations) | 3 (6) | 2 (2) | 3 (3) | 8 (9)
Neutrophil count decreased (Investigations) | 3 (8) | 3 (7) | 2 (2) | 7 (9)
Platelet count decreased (Investigations) | 1 (1) | 3 (3) | 5 (9) | 3 (5)
White blood cell count decreased (Investigations) | 4 (15) | 5 (16) | 1 (2) | 7 (12)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 5 (5) | 5 (5)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2) | 1 (1) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6) | 2 (2) | 2 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 3 (4) | 3 (6)
Bone pain (Musculoskeletal and connective tissue disorders) | 10 (13) | 11 (16) | 9 (13) | 7 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 8 (11) | 13 (17) | 4 (9) | 5 (13)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 6 (7) | 3 (3) | 6 (8)
Dysgeusia (Nervous system disorders) | 2 (3) | 6 (7) | 3 (3) | 4 (7)
Headache (Nervous system disorders) | 1 (1) | 8 (10) | 7 (8) | 6 (7)
Neuropathy peripheral (Nervous system disorders) | 2 (2) | 4 (5) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 4 (5) | 13 (13) | 8 (11) | 8 (9)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (3) | 8 (11) | 0 (0) | 6 (8)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2) | 1 (1) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (5) | 4 (6) | 6 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 3 (6) | 7 (10)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 4 (7) | 2 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 22 (22) | 18 (18) | 14 (15) | 16 (16)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (6) | 3 (5) | 1 (3)
Nail disorder (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 5 (5) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 6 (6) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 6 (7) | 5 (6) | 3 (3) | 8 (13)
Phlebitis (Vascular disorders) | 2 (3) | 1 (1) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days